CLINICAL TRIAL: NCT06617546
Title: A Randomized, Double-Blind, Placebo-Controlled, First-in-Human Study to Assess Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single and Multiple Ascending Doses of FTX-101 After Subcutaneous Injection of FTX-101 in Healthy Male Subjects
Brief Title: SAD and MAD Study of FTX-101 in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study's goals have been achieved based on a preliminary analysis of available pharmacokinetic and safety data, which demonstrate that sufficient information has been obtained.
Sponsor: Find Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FTX0101
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: remyelination; myelin; plexin A1; neuropilin 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A (SAD): Cohort A1 (Experimental): Single dose (as 1, 2 or 4 SC injection[s]) of FTX-101 or placebo in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part A (SAD): Cohort A2 (Experimental): Single dose (as 1, 2 or 4 SC injection[s]) of FTX-101 or placebo in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part A (SAD): Cohort A3 (Experimental): Single dose (as 1, 2 or 4 SC injection[s]) of FTX-101 or placebo in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part A (SAD): Cohort A4 (Experimental): Single dose (as 1, 2 or 4 SC injection[s]) of FTX-101 or placebo in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part A (SAD): Cohort A5 (Experimental): Single dose (as 1, 2 or 4 SC injection[s]) of FTX-101 or placebo in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part A (SAD): Cohort A6 (Experimental): Optional cohort to receive additional single ascending intermediate (lower) or equivalent dose (as 1, 2 or 4 SC injection[s]) of FTX-101 or placebo in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part B (MAD): Cohort B1 (Experimental): Once daily dose (as 1 or 2 SC injection[s]) of FTX-101 or placebo for 14 days in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part B (MAD): Cohort B2 (Experimental): Once daily dose (as 1 or 2 SC injection[s]) of FTX-101 or placebo for 14 days in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part B (MAD): Cohort B3 (Experimental): Once daily dose (as 1 or 2 SC injection[s]) of FTX-101 or placebo for 14 days in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo
- Part B (MAD): Cohort B4 (Experimental): Optional cohort to receive once daily dose (as 1 or 2 SC injection[s]) of FTX-101 or placebo for 14 days in a 3:1 ratio
  Interventions: Drug: FTX-101; Drug: Placebo

INTERVENTIONS:
Drug: FTX-101 — Lyophilized powder for subcutaneous injection
Drug: Placebo — Lyophilized powder for subcutaneous injection

SUMMARY:
This is a Phase 1, first-in-human (FIH), single-center, randomized, double-blind, placebo-controlled study in healthy male subjects. The study will include the following 2 parts:

* Part A: Single Ascending Dose (SAD) in healthy male subjects
* Part B: Multiple Ascending Dose (MAD) in healthy male subjects

DETAILED DESCRIPTION:
Study Rationale:

FTX-101 is a first-in-class, synthetic peptide with a novel mechanism of action designed to promote the self-repair of myelin. FTX-101 is a highly selective modulator of the PlexinA1/Neuropilin 1 receptor system and displays no significant activity on any other target. FTX-101 interferes with the heterodimerization of the coreceptor system and, ultimately, with the activation of second messenger signaling pathways shown to inhibit both the differentiation and migration of oligodendrocyte precursor cells (OPCs) and oligodendrocytes (OLs). Through this mechanism, FTX-101 disinhibits both the differentiation of OPCs to OLs and migration of OPCs into lesions, favorably promoting the remyelination process. The study is designed to evaluate the safety, tolerability and pharmacokinetic profile of single ascending doses and multiple ascending doses of FTX-101 subcutaneous injection in healthy male subjects. The study will characterize the pharmacokinetics of FTX-101 following SAD and MAD SC injection of FTX-101. The study will also evaluate the immunogenic potential of FTX-101 and will also explore the relationship between FTX-101 concentration and the change from baseline corrected QT interval.

Detailed Description:

This is a Phase 1, first-in-human (FIH), single-center, randomized, double-blind, placebo-controlled study in healthy male subjects. The study will include the following 2 parts:

* Part A: SAD in healthy male subjects
* Part B: MAD in healthy male subjects

Part A - SAD:

Part A consists of 5 planned cohorts (A1 to A5) of 8 healthy adult male subjects each. An additional SAD intermediate (lower) or equivalent dose cohort (A6) of 8 male subjects may be added at the discretion of the Sponsor. In each cohort, subjects will be randomized to receive a single subcutaneous (SC) dose (as 1, 2 or 4 injection[s]) of either FTX-101 or placebo in a 3:1 (FTX-101: placebo) ratio to have a total of 6 subjects receiving FTX-101 and 2 subjects receiving placebo.

Part B - MAD:

Part B consists of 3 planned cohorts (B1 to B3) of 8 healthy adult male subjects each. An additional MAD cohort (B4) of 8 male subjects may be added at the discretion of the Sponsor depending on emerging safety and plasma PK data from the previous cohort(s). The proposed dosing regimen (dose level and frequency) for the first cohort (B1) in Part B (MAD) will be based on available safety, tolerability, and PK data from Part A (SAD). The dosing regimens for each subsequent cohort in Part B will be determined based on the available blinded safety, tolerability, and PK data from Part A and any previous cohorts in Part B. In each cohort, subjects will be randomized to receive multiple SC doses of either FTX-101 or placebo in a 3:1 (FTX-101: placebo) ratio to have a total of 6 subjects receiving FTX-101 and 2 subjects receiving placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Willingness to comply with all study procedures and availability for the duration of the study
* Healthy adult male
* Aged at least 18 years but not older than 59 years
* Body mass index (BMI) within 18.5 kg/m^2 to 32.0 kg/m^2, inclusively
* Non- or ex-smoker
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG.

Key Exclusion Criteria:

* Supine or semi-supine pulse rate less than 45 beats per minute (bpm) or more than 100 bpm
* Supine or semi-supine blood pressure below 90/50 mmHg
* Supine or semi-supine blood pressure higher than 150/95 mmHg
* History of significant hypersensitivity to FTX-101 or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability
* History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* Showing suicidal tendency from 6 months prior to screening
* Presence of out-of-range cardiac intervals at screening defined as:

  * PR < 110 msec, PR > 200 msec
  * QRS < 60 msec, QRS >110 msec)
  * QT Interval Corrected for Heart Rate using Fridericia's Correction Formula (QTcF): • > 450 msec
  * History of additional risk factors for torsade's de pointes
  * Use of concomitant medications that prolong the QT/ corrected QT (QTc) interval
* Current use (in the last 6 months) of alcohol (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any history of substance or alcohol use disorder within the past 2 years and/or current maintenance therapy (within the past 2 years) for treatment of substance use disorder
* Use of any prescription drugs in the 28 days or 5 half-lives, whichever is longer, prior to the first study treatment administration, that in the opinion of an investigator would put into question the status of the participant as healthy
* Use of St. John's wort in the 28 days prior to the first study treatment administration
* Positive screening results to HIV Ag/Ab combo, hepatitis B surface Ag or hepatitis C virus tests
* Intake of an investigational product (IP) in the 28 days prior to the first study treatment administration or within 5 times the elimination half-life of the IP, whichever is longer
* Donation of plasma in the 7 days prior to the first study treatment administration
* Donation of 1 unit of blood to American Red Cross or equivalent organization or donation of over 500 mL of blood in the 56 days prior to the first study treatment administration

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | Part A (SAD): Days -1-15; Part B (MAD): Days -1-28
  Frequency of AE will be collected through AE monitoring.
Severity of adverse events | Part A (SAD): Days -1-15; Part B (MAD): Days -1-28
  Severity of AE will be collected through AE monitoring. AEs will be graded per the current National Cancer Institute's Common Terminology Criteria for Adverse Events.
Number of patients with a change in general biochemistry, hematology, coagulation and urinalysis clinical laboratory parameters | Part A (SAD): Days -1, 4 and 15; Part B (MAD): Days -1, 5, 9, 13, 17, 28
  Frequency of abnormal general biochemistry, hematology, coagulation, and urinalysis clinical laboratory values.
Number of patients with a change in vital signs | Part A (SAD): Days -1-4 and 15; Part B (MAD): Days -1-17 and 28
  Frequency of abnormal vital sign measurements.
Number of patients with a change in 12-lead safety electrocardiogram (ECG) | Part A (SAD): Days -1-2, and 15; Part B (MAD): Days -1, 1, 3, 5, 7, 9, 11, 14, 28
  Frequency of abnormal 12-lead ECG parameters including PR, RR, QRS, QT and QTcF.
Number of patients with a change in physical examination findings | Part A (SAD): Days -1-4, and 15; Part B (MAD): Days -1-17, 28
  Frequency of abnormal physical examination findings.
Number of patients with a change in neurological examination findings | Part A (SAD): Days 1, 2, 4, and 15; Part B (MAD): Days 1, 2, 5, 9, 14, 15, 17, and 29
  Frequency of abnormal neurological examination findings.
Frequency of injection site reactions | Part A (SAD): Days 1, 2, and 15; Part B (MAD): Days 1-14, and 28
  Evaluation of pain, tenderness, erythema/redness, swelling/induration or itching at the injection site will be rated mild (Grade 1), moderate (Grade 2), Severe (Grade 3), or potentially life-threatening (Grade 4)
Change in Columbia Suicide Severity Rating Scale (C-SSRS) score | Part A (SAD): Days -1-4, and 15; Part B (MAD:) Days -1-17, and 28
  Frequency of positive results for suicidality. The C-SSRS is a questionnaire designed for the assessment of suicidal ideation and behavior in adolescents and adults.

SECONDARY OUTCOMES:
Plasma Cmax | Part A (SAD): Days 1-4; Part B (MAD): Days 1-2
  Peak or maximum observed concentration
Plasma Tmax | Part A (SAD): Days 1-4; Part B (MAD): Days 1-2
  Time of maximum observed concentration. If the maximum observed concentration is not unique, then the first maximum is used
Plasma AUC0-last | Part A (SAD): Days 1-4; Part B (MAD): Days 1-2
  Area under the concentration-time curve from dosing to the time of last quantifiable concentration (Tlast)
Plasma AUC0-∞ (Part A) | Part A (SAD): Days 1-4
  Area under the concentration time curve extrapolated to infinity, calculated as AUClast + Clast/λZ, where Clast is the last quantifiable concentration at time Tlast
Plasma AUC0-last/∞ (Part A) | Part A (SAD): Days 1-4
  Relative percentage of AUC0-last with respect to AUC0-∞
Plasma λz | Part A (SAD): Days 1-4; Part B (MAD): Day 14-17
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus the time curve
Plasma CL/F (Part A) | Part A (SAD): Days 1-4
  Apparent clearance, calculated as Dose/AUC0-∞
Plasma Vz/F (Part A) | Part A (SAD): Days 1-4
  Apparent volume of distribution, calculated as Dose/ λZ * AUC0-∞
Plasma Thalf (Part A) | Part A (SAD): Days 1-4
  Terminal elimination half-life, calculated as ln (2)/λZ
Plasma Cmax/D (Part A) | Part A (SAD): Days 1-4
  Dose-normalized Cmax, calculated as Cmax/dose
Plasma AUC0-last/D (Part A) | Part A (SAD): Days 1-4
  Dose-normalized AUC0-last, calculated as AUC0-last/dose
Plasma AUC0-∞/D (Part A) | Part A (SAD): Days 1-4
  Dose normalized AUC 0-∞, calculated as AUC0-∞/dose
Plasma AUMC0-last (Part A) | Part A (SAD): Days 1-4
  Area under the moment curve (AUMC) from the time of dosing to the last measurable (positive) concentration
Plasma AUMC∞ (Part A) | Part A (SAD): Days 1-4
  AUMC extrapolated to infinity, based on the last observed concentration
Plasma AUC0-24 (Part B MAD) | Days 1-2
  Area under the concentration-time curve over the dosing interval
Plasma Ctrough (Part B MAD) | Days 11 to 13
  Plasma trough observed concentrations, for Day 11 to Day 13
Plasma Cmin,ss (Part B MAD) | Days 14-17
  Minimum observed concentration at steady state
Plasma Cmax,ss (Part B MAD) | Days 14-17
  Peak or maximum observed concentration at steady state
Plasma AUC0-τ (Part B MAD) | Days 14-17
  Area under the concentration-time curve over the dosing interval
Plasma Tmax,ss (Part B MAD) | Days 14-17
  Time of maximum observed concentration at steady state
Plasma Thalf (Part B MAD) | Days 14-17
  Terminal elimination half-life, calculated as ln(2)/λZ
Plasma Cav (Part B MAD) | Days 14-17
  Average steady-state plasma drug concentration calculated as AUC0-τ/τ
Plasma Fluctuation (Part B MAD) | Days 14-17
  The range of steady-state concentrations divided by the average concentration (Day 14 only)
Plasma Swing (Part B MAD) | Days 14-17
  Degree of swing over a dosing interval, after the last dose of a multiple-dose regimen expressed as a percentage. Calculated as 100*(Cmax-Cmin/Cmin).
Plasma Rac(Cmax) (Part B MAD) | Days 1-2, and 14-17
  Accumulation ratio evaluated by comparing Day 14 Cmax,ss to Day 1 Cmax
Plasma Rac(AUC) (Part B MAD) | Days 1-2, and 14-17
  Accumulation ratio evaluated by comparing Day 14 AUC0-τ to Day 1 AUC0-24
Urine Ae(0-last) | Part A (SAD): Days 1-4; Part B (MAD): Days 1, 2, and 14-17
  Cumulative amount excreted over all time intervals (0 to Tlast), calculated as the sum of all amounts excreted from each interval (t1-t2)
Urine fe | Part A (SAD): Days 1-4; Part B (MAD): Days 1, 2, and 14-17
  Fraction of unchanged drug excreted in urine during the time interval (expressed in %, calculated)
Urine CLR | Part A (SAD): Days 1-4; Part B (MAD): Days 1, 2, and 14-17
  Renal Clearance (Ae(0-last)/ AUC0-last)
Plasma CLss/F (Part B MAD) | Part B (MAD): Days 14-17
  Apparent clearance at steady state, calculated as Dose/AUC0-τ
Plasma Vz/F (Part B MAD) | Part B (MAD): Days 14-17
  Apparent volume of distribution at steady state, calculated as Dose/ λZ * AUC0-τ

CONTACTS AND LOCATIONS:
Overall Officials: Martin K. Kankam, MD, PhD, MPH, FAPCR, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No